CLINICAL TRIAL: NCT00559949
Title: Phase 2 Study of Selumetinib Hydrogen Sulfate in Iodine-131 Refractory Papillary Thyroid Carcinoma and Papillary Thyroid Carcinoma With Follicular Elements
Brief Title: Selumetinib in Treating Patients With Papillary Thyroid Cancer That Did Not Respond to Radioactive Iodine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01056; NCI-2009-01056 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LOI 7918; CDR0000574262; LOI 7918 (Other: Moffitt Cancer Center); 7918 (Other: CTEP); N01CM62201 (NIH); N01CM62203 (NIH); N01CM62208 (NIH); P30CA076292 (NIH); NCT00589940 (obsolete NCT alias)
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Recurrent Thyroid Gland Carcinoma; Stage I Thyroid Gland Papillary Carcinoma; Stage II Thyroid Gland Papillary Carcinoma; Stage III Thyroid Gland Papillary Carcinoma; Stage IV Thyroid Gland Papillary Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral selumetinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib — Selumetinib was administered orally as a free base suspension at a dose of 100 mg twice daily for 28-day cycles. Those participants experiencing Common Terminology Criteria for Adverse Events (CTCAE) v3.0 grade 3 toxicity or worse had their dose reduced to 50 mg twice daily and then to 50 mg once daily, if necessary.
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
This phase II trial is studying how well selumetinib works in treating patients with papillary thyroid cancer that did not respond to radioactive iodine. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Ascertain the objective response rate (complete response and partial response) in patients with iodine I 131-refractory papillary thyroid cancer treated with selumetinib.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this treatment in these patients. II. Determine the pharmacokinetic profile of this treatment in these patients. III. Determine the progression-free and overall survival of these patients. IV. Assess proxy measures of treatment response (thyroglobulin and PET scan) in patients treated with selumetinib.

IV. Compare relevant laboratory correlates between responders and non-responders.

OUTLINE: This is a multicenter study.

Patients receive oral selumetinib twice daily on days 1-28. Treatment repeats every 28 days in the absence of unacceptable toxicity or disease progression.

Archived tissue is examined for gene mutations, including RET, BRAF, NTRK, and RAS, by fluorescence in situ hybridization and/or polymerase chain reaction and fluorescence melting curve analysis. Protein expression of ERK and phosphorylated ERK is assessed by immunohistochemical staining.

Blood samples are collected periodically for pharmacokinetic analysis and biomarker assessment (thyroglobulin and antithyroglobulin autoantibodies).

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed papillary thyroid cancer or papillary thyroid cancer with follicular elements
* No longer amenable to radioactive iodine therapy or curative surgical resection

  * Tumor is no longer iodine avid
  * Tumor did not respond to the most recent radioactive iodine treatment
  * Patient is ineligible for further radioactive iodine therapy due to medical contraindications (e.g., lung toxicity)
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* Evidence of disease progression (objective growth of existing tumors)

  * New or enlarging measurable lesions within the past 12 months
  * If the most recent imaging study is older than 12 months, patients will still be eligible if objectively measurable disease progression is associated with clinical symptoms
* Archival tumor tissue available for mutational analysis
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* WBC ≥ 3,000/µL
* ANC ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Total bilirubin normal
* AST and ALT < 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 4 weeks after completion of study treatment
* Able to understand and willing to sign a written informed consent document
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib (AZD6244) or its excipient Captisol®
* QTc interval > 450 msec or other factors that increase the risk of QT prolongation
* Arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome), including heart failure that meets NYHA class III and IV definition
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Concurrent uncontrolled illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* At least 4 weeks since prior radiotherapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* Prior treatment with tyrosine kinase inhibitors that target RET or RAF
* Prior treatment with MEK inhibitors
* Concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent medication that can prolong the QT interval
* Other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Neil Hayes, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (6):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hayes DN, Lucas AS, Tanvetyanon T, Krzyzanowska MK, Chung CH, Murphy BA, Gilbert J, Mehra R, Moore DT, Sheikh A, Hoskins J, Hayward MC, Zhao N, O'Connor W, Weck KE, Cohen RB, Cohen EE. Phase II efficacy and pharmacogenomic study of Selumetinib (AZD6244; ARRY-142886) in iodine-131 refractory papillary thyroid carcinoma with or without follicular elements. Clin Cancer Res. 2012 Apr 1;18(7):2056-65. doi: 10.1158/1078-0432.CCR-11-0563. Epub 2012 Jan 12. PMID 22241789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 11, 2007 and June 30, 2009, 39 patients were enrolled at 5 cancer centers in the United States and one cancer center in Canada.
Period: Overall Study
Arm/Group | Arm I
Started | 39
Completed | 32
Not Completed | 7
Not completed — Progressive Disease during cycle 1 | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 4
Not completed — No disease evaluation per protocol | 1

BASELINE CHARACTERISTICS:
Population: All participants, unless specified differently in an Outcome Measure.
Arm/Group | Arm I
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 86]
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 26
Region of Enrollment [Number; unit: participants]
  Canada | 5
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR: Complete Response (CR) and Partial Response (PR) evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST). CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. A conservative estimate of the response rate of the best-studied agent in this disease, doxorubicin, is approximately 5%. Therefore, investigators will assume that selumetinib (AZD6244, NSC 741078) would be worth further pursuit if the response rate (CR+PR) were at least 20%.
Time Frame: Up to 2 years
Population: All evaluable participants
Measure: Count of Participants; unit: Participants
Groups:
- All Evaluable Participants: Participants evaluable according to protocol guidelines at time of analysis.
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 32
Participants | 1

2. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death. Progression evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST). Progressive Disease (PD): 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm. Secondary end points include toxicity, progression free survival, and overall survival. Due to the small sample size and absence of high quality historic data for this disease, these analyses were planned to be mostly exploratory and descriptive in nature.
Time Frame: Up to 2 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 39
weeks | 32 [8.4 to 56]

3. Secondary Outcome: Occurrence of Treatment Related Adverse Events
Description: Number of participants with related adverse events, per category and Grade category. Toxicity assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 2 years
Population: All participants
Measure: Number; unit: adverse events
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 39
adverse events
  Grade 1-2 - Rash | 23
  Grade 1-2 - Diarrhea | 17
  Grade 1-2 - Fatigue | 16
  Grade 1-2 - Peripheral edema | 12
  Grade 1-2 - Elevated liver enzymes | 9
  Grade 1-2 - Electrolyte abnormalities | 7
  Grade 1-2 - Nausea/vomiting | 7
  Grade 1-2 - Stomatitis | 6
  Grade 1-2 - Dyspnea | 5
  Grade 3-4 - Rash | 7
  Grade 3-4 - Diarrhea | 2
  Grade 3-4 - Fatigue | 3
  Grade 3-4 - Peripheral edema | 2
  Grade 3-4 - Elevated liver enzymes | 0
  Grade 3-4 - Electrolyte abnormalities | 0
  Grade 3-4 - Nausea/vomiting | 0
  Grade 3-4 - Stomatitis | 1
  Grade 3-4 - Dyspnea | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival using the Kaplan-Meier method with associated confidence intervals. OS analysis was intended to be mostly exploratory and descriptive in nature.
Time Frame: Up to 2 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 39
months | NA [1 to NA] — Due to the long survival time in this disease, actuarial overall survival cannot be estimated during this timeframe. High end of range has not been met.

ADVERSE EVENTS:
Time Frame: From first on treatment date to 30 days post last off treatment date, 7 years, 8 months.
Description: All participants were evaluated for adverse events.
Groups:
- All Participants: All participants on study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 7/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=39)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=39)
Anemia (Blood and lymphatic system disorders) | 10 (21)
Blurred vision (Eye disorders) | 3 (4)
Extraocular muscle paresis (Eye disorders) | 3 (3)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 21 (34)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 9 (15)
Vomiting (Gastrointestinal disorders) | 5 (6)
Fatigue (General disorders) | 24 (37)
Edema face (General disorders) | 7 (13)
Edema limbs (General disorders) | 14 (22)
Fever (General disorders) | 3 (4)
Flu like symptoms (General disorders) | 2 (5)
Pain (General disorders) | 6 (6)
Bronchial infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 5 (6)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 8 (12)
Alkaline phosphatase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 6 (10)
Creatinine increased (Investigations) | 2 (9)
Lymphocyte count decreased (Investigations) | 6 (14)
Neutrophil count decreased (Investigations) | 4 (4)
Platelet count decreased (Investigations) | 3 (4)
Weight gain (Investigations) | 4 (4)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 7 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 4 (7)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (8)
Depression (Psychiatric disorders) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 12 (27)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (33)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (9)
Thromboembolic event (Vascular disorders) | 2 (4)

LIMITATIONS AND CAVEATS:
Actuarial OS cannot be estimated due to long survival times in this disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less